CLINICAL TRIAL: NCT00005296
Title: Sleep Apnea: Age Effects On Prevalence and Natural History
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Edward Bixler, Principal Investigator, Milton S. Hershey Medical Center
Other Study IDs: 2019; R01HL040916 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify the prevalence of sleep apnea in men and its relationship to age, assess the natural history of the disorder, and predict those men at risk.

DETAILED DESCRIPTION:
BACKGROUND:

Sleep apnea is potentially a life-threatening disorder commonly associated with the aging process. Often sleep apnea is accompanied by considerable morbidity for both physical and mental health; the associated excessive daytime sleepiness, cardiovascular abnormalities, and cognitive impairment impact greatly on daytime functioning. In 1990, the prevalence of sleep apnea in the general population was undetermined, and there was much speculation regarding its natural history.

DESIGN NARRATIVE:

For the prevalence study, 4,364 randomly-sampled men selected from the general population and stratified by age were evaluated for risk factors for sleep apnea. A total of 741 men found to be at risk were evaluated in the sleep laboratory to determine the degree, if any, of sleep apnea or sleep disordered breathing. Prior to recording subjects in the sleep laboratory, a thorough history was obtained from each subject and a physical examination completed. All men entering into the first four years of the prevalence portion of the study who were found to have sleep apnea or sleep disordered breathing were reevaluated yearly over a five year period in the natural history part of the study. The natural history portion also included 150 men previously studied in the sleep laboratory for apnea but who were not part of the random sample of 4,000 and who were not part of the prevalence study.

ELIGIBILITY:
stratified random sample based on risk severity for sleep disordered breathing based on phone interview

Ages: 20 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stratified random sample following phone interview
Sampling Method: Probability Sample
Enrollment: 741 (Actual)
Dates: Start 1990-01 (Actual); Primary Completion 1995-01-18 (Actual); Study Completion 1995-01-18 (Actual)

PRIMARY OUTCOMES:
sleep disordered breathing | immediately upon time of recording
  Apnea/hypopnea index

REFERENCES:
- [Background] Bixler EO, Vgontzas AN, Ten Have T, Tyson K, Kales A. Effects of age on sleep apnea in men: I. Prevalence and severity. Am J Respir Crit Care Med. 1998 Jan;157(1):144-8. doi: 10.1164/ajrccm.157.1.9706079. PMID 9445292